CLINICAL TRIAL: NCT03292419
Title: A Prospective Evaluation of Topography-guided LASIK Surgery
Brief Title: Topography-guided LASIK Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43306
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Topography guided
Masking Description: N0ne
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topography guided LASI (Other)
  Interventions: Procedure: Topography-guided LASIK

INTERVENTIONS:
Procedure: Topography-guided LASIK — LASIK surgery

SUMMARY:
The investigators are analyzing outcomes of topography-guided LASIK surgery in participants with myopia and myopic astigmatism

DETAILED DESCRIPTION:
The investigators are analyzing outcomes of topography-guided LASIK surgery in participants with myopia and myopic astigmatism. The investigators will be monitoring changes in anterior segment optical coherence tomography epithelial thickness maps. The investigators will compare preoperative maps to postoperative maps at one, three, six and twelve months. In addition, the investigators will measure changes in epithelial maps from postoperative month through twelve months to help understand what is happening to the corneal epithelium to try to explain why UDVA and CDVA improves over time

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 and older with healthy eyes. Nearsightedness between -0.50 diopters and -8.00 diopters.
* Subjects with up to 3.00 diopters of astigmatism.
* Subjects with a spherical equivalent of up to -9.00 diopters.

Exclusion Criteria:

* Subjects under the age of 18.
* Subjects with excessively thin corneas.
* Subjects with topographic evidence of keratoconus.
* Subjects with ectatic eye disorders.
* Subjects with autoimmune diseases.
* Subjects who are pregnant or nursing.
* Subjects with more than 3.00 diopters of astigmatism

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Epithelial thickness maps | 12 months
  Changes in anterior segment optical coherence tomography epithelial thickness maps.

SECONDARY OUTCOMES:
Changes in corrected visual acuity | 12 months
  Corrected distance visual acuity (CDVA)
Uncorrected distance visual acuity | 12 months
  Uncorrected distance visual acuity (UDVA)
Quality of Vision | 12 months
  Patient reported outcomes questionnaire
Predictability | 12 months
  Percentage of eyes within +/-0.25, 0.50 and 1.00 diopter of the intended correction
Contrast visual acuity | 12 months
  5 and 25% ETDRS contrast acuity
Residual astigmatism levels after surgery | 12 months
  Vector analysis of astigmatic outcomes
Change in refraction over time | 12 months
  Change in spherical equivalent over time

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No